CLINICAL TRIAL: NCT00302718
Title: RCT of Financial Incentives to Translate ALLHAT Into Practice
Brief Title: Financial Incentives to Translate ALLHAT Into Practice: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 04-349; R01HL079173 (NIH)
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
Keywords: Physician Incentive Plan; Quality of Health Care; Reimbursement, Incentive; Randomized Controlled Trial; Physicians; Reward
MeSH Terms: conditions — Hypertension | interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Physician-level incentives (Experimental): Examines the effect of physician-level financial incentives on hypertension quality of care
  Interventions: Behavioral: Physician-level financial incentives
- Practice-level incentives (Experimental): Examines the effect of practice-level financial incentives on hypertension quality of care
  Interventions: Behavioral: Practice-level financial incentives
- Physician- and practice-level incentives (Experimental): Examines the effect of physician- and practice-level financial incentives on hypertension quality of care
  Interventions: Behavioral: Physician- and practice-level financial incentives
- No incentives (control) (No Intervention): Physician participants in this arm received only audit and feedback performance reports as did the participants in the intervention arms.

INTERVENTIONS:
Behavioral: Physician-level financial incentives — Enrolled physician participants are eligible to receive financial incentives and audit and feedback reports based on their performance during a 4-month interval on the hypertension care study outcomes.
  Arms: Physician-level incentives
Behavioral: Practice-level financial incentives — Enrolled practices (physician physicians and non-physician primary care personnel) are eligible to receive financial incentives and audit and feedback reports based on the performance of the practice during a 4-month interval on the hypertension care study outcomes.
  Arms: Practice-level incentives
Behavioral: Physician- and practice-level financial incentives — Enrolled participants are eligible to receive financial incentives and audit and feedback reports based on performance during a 4-month interval on the hypertension care study outcomes. This arm tests the effect of combined financial incentives (physician-level incentives and practice-level incentives).
  Arms: Physician- and practice-level incentives

SUMMARY:
The purpose of this study was to determine whether financial incentives for guideline-recommended treatment of hypertension are effective. We hypothesized that patients with hypertension cared for by physicians or practice groups receiving financial incentives were more likely to be prescribed guideline-recommended anti-hypertensive medications and achieve Joint National Commission (JNC) 7 guideline-recommended blood pressure goals compared to patients who were treated by providers that did not receive financial incentives.

DETAILED DESCRIPTION:
Background:

Despite compelling evidence of the benefits of treatment, hypertension is controlled in less than one-quarter of US citizens. Using a cluster randomized controlled trial, we tested the effect of explicit physician-level and practice-level financial incentives to promote the provision of guideline-recommended anti-hypertensive medications and improved control of hypertension in the VA primary care setting.

Objectives:

The goals were to: (1) determine the effect of physician-level financial incentives on processes and outcomes of care for outpatients with hypertension; (2) assess the impact of practice-level incentives; (3) ascertain whether there were additive or synergistic effects of physician- and practice-level incentives; (4) evaluate the persistence of the effect of incentives after the intervention ceases; and (5) identify any negative impacts of incentives on patients, providers, or health care organizations.

Methods:

We randomized 12 VA hospital-based outpatient clinics to the following arms: (1) physician-level incentives; (2) practice-level incentives; (3) physician- and practice-level incentives; and (4) no incentives. We enrolled 83 primary care physicians and 42 practice group members (e.g., nurses). All participants received audit and feedback performance reports. Study measures included the use of guideline-recommended anti-hypertensive medications and the proportion of patients who achieved national (JNC 7) guideline-recommended blood pressure goals or received an appropriate response to uncontrolled blood pressure. The intervention period consisted of five four-month performance periods. For each period, trained reviewers collected medications, blood pressure readings, comorbid conditions, medication allergies, and lifestyle recommendations from the VA electronic health record system for a sample of eligible patients from the physicians' panels. After the final performance report, we implemented a 12-month washout period. To determine the impact of incentives for the intervention period, we performed a repeated-measures longitudinal analysis using the hospital as a random effect. We evaluated the rate of change in the proportion of patients who met the study measures over time for the intervention group physicians. We assessed post-washout performance using a linear analysis with clustering by hospital. To evaluate unintended consequences of the incentives, we examined the incidence of hypotension in the physicians' panels.

Status:

The study is completed. The primary findings were published in September 2013 in the Journal of the American Medical Association (JAMA). We are currently preparing manuscripts describing findings from the study's secondary aims.

ELIGIBILITY:
Inclusion Criteria:

Study participants had to be full-time primary care physicians employed by the Veterans Health Administration (VA) at one of the 12 VA hospitals that participated in the study.

We defined a full-time primary care physician as spending at least 0.60 full-time equivalent (FTE) delivering patient care services in the primary care setting or having a panel size of at least 500 patients at the time of study arm randomization. The primary care settings included internal medicine, primary care medical clinics, and women's health care clinics. The trial did not actively recruit patients into the study. This study retrospectively reviewed a random sample of health records of eligible patients that had clinical encounters with the physician participants.

Exclusion Criteria:

The study did not include VA physicians that were trainees.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-02; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Petersen, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (12):
- United States (12):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - VA Connecticut Health Care System (Newington), Newington, Connecticut
  - VA Medical Center, Augusta, Augusta, Georgia
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - Aleda E. Lutz VA Medical Center, Saginaw, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, Jackson, Mississippi
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Medical Center, Providence, Providence, Rhode Island
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

REFERENCES:
- [Result] Petersen LA, Simpson K, Pietz K, Urech TH, Hysong SJ, Profit J, Conrad DA, Dudley RA, Woodard LD. Effects of individual physician-level and practice-level financial incentives on hypertension care: a randomized trial. JAMA. 2013 Sep 11;310(10):1042-50. doi: 10.1001/jama.2013.276303. PMID 24026599
- [Result] Hysong SJ, Simpson K, Pietz K, SoRelle R, Broussard Smitham K, Petersen LA. Financial incentives and physician commitment to guideline-recommended hypertension management. Am J Manag Care. 2012 Oct 1;18(10):e378-91. PMID 23145846
- [Result] Petersen LA, Woodard LD, Urech TH. Financial incentives to control hypertension in patients--reply. JAMA. 2014 Jan 15;311(3):303-4. doi: 10.1001/jama.2013.284315. No abstract available. PMID 24430324
- [Result] Woodard LD, Landrum CR, Urech TH, Wang D, Virani SS, Petersen LA. Impact of clinical complexity on the quality of diabetes care. Am J Manag Care. 2012 Sep;18(9):508-14. PMID 23009301
- [Result] Petersen LA, Simpson K, Sorelle R, Urech T, Chitwood SS. How variability in the institutional review board review process affects minimal-risk multisite health services research. Ann Intern Med. 2012 May 15;156(10):728-35. doi: 10.7326/0003-4819-156-10-201205150-00011. PMID 22586010
- [Result] Woodard LD, Urech T, Landrum CR, Wang D, Petersen LA. Impact of comorbidity type on measures of quality for diabetes care. Med Care. 2011 Jun;49(6):605-10. doi: 10.1097/MLR.0b013e31820f0ed0. PMID 21422952
- [Result] Virani SS, Steinberg L, Murray T, Negi S, Nambi V, Woodard LD, Bozkurt B, Petersen LA, Ballantyne CM. Barriers to non-HDL cholesterol goal attainment by providers. Am J Med. 2011 Sep;124(9):876-80.e2. doi: 10.1016/j.amjmed.2011.02.012. PMID 21854896
- [Result] Petersen LA, Urech T, Simpson K, Pietz K, Hysong SJ, Profit J, Conrad D, Dudley RA, Lutschg MZ, Petzel R, Woodard LD. Design, rationale, and baseline characteristics of a cluster randomized controlled trial of pay for performance for hypertension treatment: study protocol. Implement Sci. 2011 Oct 3;6:114. doi: 10.1186/1748-5908-6-114. PMID 21967830
- [Result] Petersen LA. Pay for performance in myocardial infarction: are we reaping the rewards? Nat Clin Pract Cardiovasc Med. 2008 Mar;5(3):134-5. doi: 10.1038/ncpcardio1069. Epub 2007 Dec 4. No abstract available. PMID 18059383
- [Result] Van Swol MA. Does pay-for-performance improve the quality of health care? Ann Intern Med. 2007 Apr 3;146(7):538; author reply 538-9. doi: 10.7326/0003-4819-146-7-200704030-00015. No abstract available. PMID 17404361
- [Result] Petersen LA, Urech TH, Byrne MM, Pietz K. Do financial incentives in a globally budgeted healthcare payment system produce changes in the way patients are categorized? A five-year study. Am J Manag Care. 2007 Sep;13(9):513-22. PMID 17803365
- [Result] Petersen LA, Simpson K, Urech T, Woodard L, Hysong S, Dudley RA. Do financial incentives to health care providers generate greater interest in adhering to performance measures than audit and feedback alone. Journal of general internal medicine. 2009 Apr 1; 24(S1):S58-S59.
- [Result] Petersen LA, Woodard LD, Henderson LM, Urech TH, Pietz K. Will hypertension performance measures used for pay-for-performance programs penalize those who care for medically complex patients? Circulation. 2009 Jun 16;119(23):2978-85. doi: 10.1161/CIRCULATIONAHA.108.836544. Epub 2009 Jun 1. PMID 19487595
- [Result] Woodard LD, Petersen LA. Improving the performance of performance measurement. J Gen Intern Med. 2010 Feb;25(2):100-1. doi: 10.1007/s11606-009-1198-z. No abstract available. PMID 19953336
- [Result] Petersen LA, Woodard LD, Urech T, Daw C, Sookanan S. Does pay-for-performance improve the quality of health care? Ann Intern Med. 2006 Aug 15;145(4):265-72. doi: 10.7326/0003-4819-145-4-200608150-00006. PMID 16908917
- [Result] Hysong SJ, Kell HJ, Petersen LA, Campbell BA, Trautner BW. Theory-based and evidence-based design of audit and feedback programmes: examples from two clinical intervention studies. BMJ Qual Saf. 2017 Apr;26(4):323-334. doi: 10.1136/bmjqs-2015-004796. Epub 2016 Jun 10. PMID 27288054
- [Result] Petersen LA, Ramos KS, Pietz K, Woodard LD. Impact of a Pay-for-Performance Program on Care for Black Patients with Hypertension: Important Answers in the Era of the Affordable Care Act. Health Serv Res. 2017 Jun;52(3):1138-1155. doi: 10.1111/1475-6773.12517. Epub 2016 Jun 22. PMID 27329344
- [Result] Hysong SJ, SoRelle R, Broussard Smitham K, Petersen LA. Reports of unintended consequences of financial incentives to improve management of hypertension. PLoS One. 2017 Sep 21;12(9):e0184856. doi: 10.1371/journal.pone.0184856. eCollection 2017. PMID 28934258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled non-physician primary care personnel at the hospitals randomized to the two study arms that tested the effect of practice-level incentives. Only data from physicians were used to assess both physician-level and practice-level performances. This participant enrollment table does not include data on the non-physician participants.
Groups:
- Physician-level Incentives: Examines the effect of physician-level financial incentives on hypertension quality of care
  Physician-level financial incentives: Enrolled physician participants were eligible to receive financial incentives based on their performance during a 4-month interval on the hypertension care study outcomes.
- Practice-level Incentives: Examines the effect of practice-level financial incentives on hypertension quality of care
  Practice-level financial incentives: Enrolled practices (physician participants and non-physician primary care personnel) were eligible to receive financial incentives based on the performance of the practice during a 4-month interval on the hypertension care study outcomes.
- Physician- and Practice-level Incentives: Examines the effect of physician and practice-level financial incentives on hypertension quality of care
  Physician- and practice-level financial incentives: Enrolled subjects were eligible to receive financial incentives based on performance during a 4-month interval on the hypertension care study outcomes. This arm tested the effect of combined financial incentives.
- No Incentives (Control): Physician participants in the control group did not receive any financial incentives. They received audit and feedback performance reports at the end of each performance period like the intervention groups.
Period: Overall Study
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Started | 20 | 21 | 21 | 21
Completed | 19 | 20 | 19 | 19
Not Completed | 1 | 1 | 2 | 2
Not completed — Participant left the hospital | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Participant left primary care setting | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Distribution of Physician Characteristics Across Study Groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control) | Total
Number analyzed (Participants) | 19 | 20 | 19 | 19 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] — One physician participant in the physician-level incentive arm declined to provide age data.
  years | 45 (8) | 48 (8) | 44 (6) | 48 (7) | 46 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 6 | 34
  Male | 8 | 12 | 10 | 13 | 43
Race/Ethnicity, Customized [Number; unit: participants] — These data describe the race of the physician participants.
  participants
    White | 7 | 7 | 9 | 8 | 31
    Black | 3 | 2 | 1 | 0 | 6
    Asian Indian | 5 | 5 | 6 | 5 | 21
    Other | 4 | 6 | 3 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 19 | 19 | 77

OUTCOME MEASURES:

1. Primary Outcome: Proportion of the Physicians' Patients With Blood Pressure Control or Appropriate Response to Uncontrolled Blood Pressure
Description: This measure reports the unadjusted proportion of physicians' patients meeting the study outcome for the first performance period (baseline). Data are based on review of the electronic health records for 40 patients with hypertension randomly selected from each physician's panel. We used the guidelines from the "Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7)" to determine if the physicians' patients achieved the recommended blood pressures thresholds and if providers appropriately responded to uncontrolled blood pressure. Appropriate responses included increasing the dosage of a guideline-recommended antihypertensive medication or recommending a lifestyle modification to patient with Stage 1 hypertension.
Time Frame: Baseline period (August-November 2007)
Population: The number of physicians listed is those who participated in the baseline period. The participant flow diagram describes the final number of physicians who received at least two instances of the intervention and were included in the repeated-measures longitudinal analysis.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: Patient records
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Number analyzed (Participants) | 19 | 18 | 17 | 18
Number analyzed (Patient records) | 760 | 720 | 680 | 720
percentage of physicians' patients | 75 | 80 | 79 | 86

2. Primary Outcome: Proportion of Physicians' Patients With Blood Pressure Control or Appropriate Response to Uncontrolled Blood Pressure
Description: This measure reports the unadjusted proportion of physicians' patients meeting the study outcome for the fifth and final intervention performance period. Data are based on review of the electronic health records for 40 patients with hypertension randomly selected from each physician's panel. We used the guidelines from the "Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7)" to determine if the physicians' patients achieved the recommended blood pressures thresholds and if providers appropriately responded to uncontrolled blood pressure. Appropriate responses included increasing the dosage of a guideline-recommended antihypertensive medication or recommending a lifestyle modification to patient with Stage 1 hypertension.
Time Frame: Final intervention period (April-July 2009)
Population: The number of physicians listed is those who participated in the final intervention period. The participant flow diagram describes the final number of physicians who received at least two instances of the intervention and were included in the repeated-measures longitudinal analysis.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: Patient records
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Number analyzed (Participants) | 18 | 19 | 15 | 19
Number analyzed (Patient records) | 720 | 760 | 600 | 760
percentage of physicians' patients | 84 | 85 | 88 | 86

3. Primary Outcome: Proportion of Physicians' Patients With Blood Pressure Control or Appropriate Response to Uncontrolled Blood Pressure
Description: This measure reports the unadjusted proportion of physicians' patients meeting the study outcome for the post-washout performance period. Data are based on review of the electronic health records for 40 patients with hypertension randomly selected from each physician's panel. We used the guidelines from the "Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7)" to determine if the physicians' patients achieved the recommended blood pressures thresholds and if providers appropriately responded to uncontrolled blood pressure. Appropriate responses included increasing the dosage of a guideline-recommended antihypertensive medication or recommending a lifestyle modification to patient with Stage 1 hypertension.
Time Frame: After the washout period (May-August 2011)
Population: The number of physicians listed is those who participated in the post-washout performance period. The participant flow diagram describes the final number of physicians who received at least two instances of the intervention and were included in the repeated-measures longitudinal analysis.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: Patient records
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Number analyzed (Participants) | 13 | 17 | 11 | 14
Number analyzed (Patient records) | 520 | 680 | 440 | 560
percentage of physicians' patients | 83 | 82 | 83 | 87

4. Primary Outcome: Proportion of Physicians' Patients Prescribed Guideline-recommended Antihypertensive Medications
Description: This measure reports the unadjusted proportion of physicians' patients meeting the study outcome for the first performance period (baseline). Data are based on review of the electronic health records for 40 patients with hypertension randomly selected from each physician's panel. We used the "Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7)" to evaluate use of guideline-recommended antihypertensive medications. Assessing use of guideline-recommended medications included collecting information about the patient's compelling conditions (e.g., diabetes mellitus) as well as allergies and refusals to antihypertensive medications.
Time Frame: Baseline period (August-November 2007)
Population: as for outcome 1
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: Patient records
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Number analyzed (Participants) | 19 | 18 | 17 | 18
Number analyzed (Patient records) | 760 | 720 | 680 | 720
percentage of physicians' patients | 61 | 56 | 65 | 63

5. Primary Outcome: Proportion of Physicians' Patients Prescribed Guideline-recommended Antihypertensive Medications
Description: This measure reports the unadjusted proportion of physicians' patients meeting the study outcome for the fifth and final intervention performance period. Data are based on review of the electronic health records for 40 patients with hypertension randomly selected from each physician's panel. We used the "Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7)" to evaluate use of guideline-recommended antihypertensive medications. Assessing use of guideline-recommended medications included collecting information about the patient's compelling conditions (e.g., diabetes mellitus) as well as allergies and refusals to antihypertensive medications.
Time Frame: Final intervention period (April-July 2009)
Population: The number of physicians listed is those who participated in the final intervention performance period. The participant flow diagram describes the final number of physicians who received at least two instances of the intervention and were included in the repeated-measures longitudinal analysis.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: Patient records
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Number analyzed (Participants) | 18 | 19 | 15 | 19
Number analyzed (Patient records) | 720 | 760 | 600 | 760
percentage of physicians' patients | 73 | 65 | 80 | 72

6. Primary Outcome: Proportion of Physicians' Patients Prescribed Guideline-recommended Antihypertensive Medications
Description: This measure reports the unadjusted proportion of physicians' patients meeting the study outcome for the post-washout performance period. Data are based on review of the electronic health records for 40 patients with hypertension randomly selected from each physician's panel. We used the "Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7)" to evaluate use of guideline-recommended antihypertensive medications. Assessing use of guideline-recommended medications included collecting information about the patient's compelling conditions (e.g., diabetes mellitus) as well as allergies and refusals to antihypertensive medications.
Time Frame: After the washout period (May-August 2011)
Population: as for outcome 3
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: Patient records
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Number analyzed (Participants) | 13 | 17 | 11 | 14
Number analyzed (Patient records) | 520 | 680 | 440 | 560
percentage of physicians' patients | 66 | 65 | 73 | 71

7. Secondary Outcome: Colorectal Cancer (CRC) Screening
Description: This measure reports the proportion of patients who had at least one of four CRC screens in the appropriate timeframe for the first performance period (baseline). Appropriate CRC screens consisted of at least one of the following: 1) fecal occult blood test every year; 2) barium enema every five years; 3) flexible sigmoidoscopy every five years; 4) colonoscopy every ten years. We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Baseline period (August - November 2007)
Population: All patients aged 51-74 at the time of qualifying visit with no history of CRC. We used data from chart reviews to evaluate this measure.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 440 | 444 | 463 | 343
percentage of physicians' patients | 80.68 | 80.18 | 79.05 | 80.47

8. Post Hoc Outcome: Incidence of Hypotension Among All Patients With Hypertension
Description: Patients had at least one primary care encounter during the interval assessed. We looked four months from the encounter for evidence of hypotension, either an outpatient systolic blood pressure (BP) < 90 mm Hg, an outpatient diagnosis of hypotension, or both.
Time Frame: Intervention period (February-May 2009)
Population: All patients with hypertension from the physicians' panel who had an outpatient encounter between February and May 2009. We used data from automated processing of structured fields from electronic health records to evaluate this measure.
Measure: Number; unit: percentage of all hypertensive patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 19 | 20 | 19
Number analyzed (patient records) | 3792 | 4677 | 4712 | 4821
percentage of all hypertensive patients | 1.4 | 1.20 | 1.15 | 1.12

9. Secondary Outcome: Colorectal Cancer (CRC) Screening
Description: This measure reports the proportion of patients who had at least one of four CRC screens in the appropriate timeframe for the fifth and final intervention performance period. Appropriate CRC screens consisted of at least one of the following: 1) fecal occult blood test every year; 2) barium enema every five years; 3) flexible sigmoidoscopy every five years; 4) colonoscopy every ten years. We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Final intervention period (April-July 2009)
Population: as for outcome 7
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 460 | 450 | 487 | 370
percentage of physicians' patients | 80.43 | 80.22 | 72.28 | 85.41
Statistical Analysis 1: Comparison: No Incentives (Control) vs Physician-level Incentives vs Practice-level Incentives vs Physician- and Practice-level Incentives; Test type: Other; p < .0001, Chi-squared

10. Secondary Outcome: Low-density Lipoprotein (LDL) Cholesterol Levels
Description: This measure reports the proportion of patients who had LDL control (LDL cholesterol < 100) for the first performance period (baseline). We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Baseline period (August-November 2007)
Population: All patients at high risk for elevated LDL. These patients have any of the following: 1) a history of ischemic heart disease, angioplasty, or coronary artery bypass grafting; 2) a history or diagnosis of peripheral artery disease or aortic aneurism; 3) a compelling indication of diabetes. We used data from chart reviews to evaluate this measure.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 374 | 355 | 365 | 326
percentage of physicians' patients | 64.17 | 66.76 | 66.58 | 68.10

11. Secondary Outcome: Low-density Lipoprotein (LDL) Cholesterol Levels
Description: This measure reports the proportion of patients who had LDL control (LDL cholesterol < 100) for the fifth and final intervention performance period. We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Final intervention period (April-July 2009)
Population: as for outcome 10
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Groups:
- Physician- and Practice- Level Incentives: Examines the effect of physician and practice-level financial incentives on hypertension quality of care Physician- and practice-level financial incentives: Enrolled subjects were eligible to receive financial incentives based on performance during a 4-month interval on the hypertension care study outcomes. This arm tested the effect of combined financial incentives.
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice- Level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 413 | 351 | 381 | 340
percentage of physicians' patients | 75.30 | 70.37 | 69.55 | 74.12
Statistical Analysis 1: Comparison: No Incentives (Control) vs Physician-level Incentives vs Practice-level Incentives vs Physician- and Practice- Level Incentives; Test type: Other; p = 0.2114, Chi-squared

12. Secondary Outcome: Hemoglobin (Hb) A1c Levels
Description: This measure reports the proportion of patients with (Hb)A1c control ((Hb)A1c ≤ 9%) for the first performance period (baseline). We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Baseline period (August-November 2007)
Population: All patients with a compelling indication of diabetes, including a history of diagnosis of diabetes, was taking diabetes medications at index visit, or has a fasting blood sugar level ≥ 126 or random blood sugar ≥ 200. We used data from chart reviews to evaluate this measure.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 238 | 271 | 270 | 217
percentage of physicians' patients | 92.02 | 90.04 | 89.63 | 91.24

13. Secondary Outcome: Hemoglobin (Hb) A1c Levels
Description: This measure reports the proportion of patients with (Hb)A1c control ((Hb)A1c ≤ 9%) for the fifth and final intervention performance period. We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Final intervention period (April-July 2009)
Population: as for outcome 12
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 283 | 243 | 265 | 235
percentage of physicians' patients | 89.05 | 91.77 | 90.94 | 91.49
Statistical Analysis 1: Comparison: No Incentives (Control) vs Physician-level Incentives vs Practice-level Incentives vs Physician- and Practice-level Incentives; Test type: Other; p = 0.6954, Chi-squared

14. Secondary Outcome: Beta Blocker Use
Description: This measure reports the proportion of patients with beta blocker use at the time of the index visit for the first performance period (baseline). We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant.
Time Frame: Baseline period (August - November 2007)
Population: All patients with at least one of the following: 1) a history of diagnosis of ischemic heart disease (IHD), angioplasty, or CABG; 2) a history of myocardial infarction (MI); 3) patients who have a history of USA. We used data from chart reviews to evaluate this measure.
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 203 | 135 | 173 | 165
percentage of physicians' patients | 60.10 | 65.93 | 64.16 | 64.24

15. Secondary Outcome: Beta Blocker Use
Description: This measure reports the proportion of patients with beta blocker use at the time of the index visit for the fifth and final intervention performance period. We did not measure the pre-specified post washout period results for this secondary outcome. The pre-specified post washout period results were not to be measured if the final intervention period results were not significant
Time Frame: Final intervention period (April-July 2009)
Population: as for outcome 14
Measure: Number; unit: percentage of physicians' patients
Units Other Than Participants: patient records
Arm/Group | No Incentives (Control) | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives
Number analyzed (Participants) | 19 | 18 | 19 | 15
Number analyzed (patient records) | 217 | 207 | 200 | 164
percentage of physicians' patients | 70.51 | 71.01 | 69.50 | 70.12
Statistical Analysis 1: Comparison: No Incentives (Control) vs Physician-level Incentives vs Practice-level Incentives vs Physician- and Practice-level Incentives; Test type: Other; p = 0.9895, Chi-squared

ADVERSE EVENTS:
Arm/Group | Physician-level Incentives | Practice-level Incentives | Physician- and Practice-level Incentives | No Incentives (Control)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes